CLINICAL TRIAL: NCT02821286
Title: Identification of Anaphylactogenic Antibodies in the Blood of Peanut Allergic Patients
Brief Title: Identification of Anaphylactogenic Antibodies in Peanut Allergy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Collaborators: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: UZH
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational study — Blood sampling

SUMMARY:
This project intends the analysis and profiling of specific antibodies against major peanut allergens in peanut allergic individuals and molecular cloning of human antibodies against major peanut allergens.

DETAILED DESCRIPTION:
* Characterization of patient samples reactivity (sera obtained from blood) against major peanut allergens.
* Isolation of antibody-producing B cells.
* Molecular cloning of peanut-specific antibodies from antibody gene sequences obtained from B cells.
* Biophysical and functional characterization of isolated antibodies

ELIGIBILITY:
Inclusion Criteria:

* Participants have a described clinical history of peanut allergy and/or are sensitized to peanut allergens (as evidenced by positive skin prick test and allergen-specific IgE testing)
* Male and female subjects older than 3 years
* Written informed consent

Exclusion Criteria:

* age below three years
* patients suffering from any disease where blood withdrawals might impact the patients' health status such as known anemia.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The project population includes patients of at least three years of age with a described history of peanut allergy and/or sensitization to peanut allergens (as evidenced by positive skin prick test or allergen-specific IgE testing).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Analysis and profiling of specific antibodies against major peanut allergens in samples derived from peanut allergic patients. | June 2016 to May 2018

IPD SHARING:
Plan to Share IPD: No